CLINICAL TRIAL: NCT07361731
Title: Evaluating the Feasibility, Acceptability, and Preliminary Outcomes of Heart Rate Variability Biofeedback for Individuals With Opioid Use Disorder.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Sunny Wonsun Kim, Ph.D, Associate Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022883
Record Dates: First submitted 2025-12-20; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Autonomic Nervous System Imbalance; Heart Rate Variability (HRV); Opioid Use Disorder; Breathing Techniques; Opioid Craving; Recovery; Emotional Regulation; Positive and Negative Affect; Stress; Biofeedback
Keywords: heart rate variability biofeedback; app based intervention; opioid use disorder; adjunct intervention; opioid cravings; daily diary
MeSH Terms: conditions — Opioid-Related Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRVB Intervention group (Experimental)
  Interventions: Behavioral: Heart rate variability biofeedback

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback — Participants non-randomized to the single intervention arm will receive a standardized HRV sensor and accompanying smartphone application, along with a 30-45-minute HRVB training session focused on using biofeedback signals to generate a resonant frequency pattern of HRV (coherence) following baseline data collection. Participants will be asked to practice their HRVB skills at home for 10 minutes per day over a 3-week period.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, acceptability, and preliminary outcomes of a heart rate variability biofeedback (HRVB) intervention among adults with opioid use disorder (OUD) receiving residential treatment. The study aims to learn whether HRVB can be implemented successfully in this setting and whether it may help participants manage stress, emotional regulation, and cravings.

The main questions this study aims to answer are:

Is HRVB feasible and acceptable for adults with OUD in a residential treatment program, as indicated by recruitment, retention, adherence, and participant satisfaction?

Do participants show preliminary improvements in stress, affect, emotional regulation, self-efficacy, and cravings following participation in the HRVB intervention?

Participants will be adults with OUD enrolled in a residential treatment program.

Participants will:

1. Complete baseline and post-intervention questionnaires assessing stress, affect, emotional regulation, social support, self-efficacy, and cravings
2. Participate in daily HRVB practice using a portable biofeedback device for approximately 3 weeks
3. Complete brief daily diary assessments related to mood, stress, and cravings

This is a single-arm pilot study designed to inform the feasibility and future refinement of HRVB as an adjunct intervention for individuals with OUD in residential treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are

  1. adults aged 18 to 65,
  2. currently admitted to a transitional living program for opioid use and within the first 30 days of admission
  3. voluntarily agree to participate and demonstrate adequate decision-making capacity as determined by the study team during informed consent
  4. able to read and speak English,
  5. have a clinical diagnosis of OUD at any severity level, whether mild, moderate, or severe,
  6. identify opioids as their primary drug of choice
  7. should have access to smartphones for daily individual practice of the intervention.
  8. must reside at the treatment program for the duration of the study

Exclusion Criteria:

1. inability to provide informed consent,
2. inability to demonstrate adequate decision-making capacity
3. currently having suicidal thoughts or psychotic symptoms
4. history of receiving previous HRVB training,
5. have a serious cardiac condition such as having pacemaker, heart failure or cardiac arrhythmia),
6. a known self-reported diagnosis of dementia, a severe brain injury, or a serious neurological condition(e.g., Parkinson's disease)
7. currently enrolled in any other biofeedback program simultaneously
8. currently taking medications such as MAOIs and alpha/beta blockers or benzodiazepines.

Participant recruitment will be conducted at the recruitment site. Individuals younger than 18 or older than 65 years are excluded from participation primarily due to age-related differences in autonomic function and heart rate variability (HRV) regulation. Restricting the sample to adults aged 18-65 allows for more accurate measurement and interpretation of HRV data, thereby reducing potential confounding effects related to age-related physiological differences.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Feasibility) | From study launch through completion of recruitment
  Recruitment feasibility will be assessed as the proportion of eligible individuals who enroll in the HRVB intervention during the recruitment period in the transitional residential treatment setting.
  Metric: Number of participants enrolled ÷ number of eligible individuals Unit of Measure: Percentage (%) of eligible individuals enrolled Benchmark: ≥ 60% enrollment of eligible individuals
Retention Rate (Feasibility) | Time Frame: From enrollment through completion of the 3-week intervention
  Description: Retention feasibility will be assessed as the proportion of enrolled participants who complete post-intervention (T2) assessments at the end of the 3-week HRVB intervention.
  Metric: Number of participants completing T2 ÷ number of participants enrolled Unit of Measure: Percentage (%) of enrolled participants completing T2 Benchmark: ≥ 80% completion of post-intervention assessments
HRVB Practice Adherence (Feasibility) | From enrollment through completion of the 3-week intervention
  Description: Adherence feasibility will be assessed as the proportion of participants who engage in consistent daily HRVB practice across the intervention period. Self-reported adherence will be corroborated using HeartCloud device data.
  Metric: Number of participants practicing on ≥70% of intervention days ÷ total number of participants Unit of Measure: Percentage (%) of participants meeting adherence threshold Benchmark: ≥ 70% of participants practice on ≥70% of intervention days
Daily Diary Compliance (Feasibility) | From enrollment through completion of the 3-week intervention
  Description: Daily diary compliance will be assessed as the proportion of expected ecological momentary assessment (EMA) diary entries completed during the intervention period.
  Metric: Number of completed diary entries ÷ number of expected diary entries Unit of Measure: Percentage (%) of expected diary entries completed Benchmark: ≥ 80% of daily diary entries completed
Intervention Acceptability Rating (Acceptability) | At the post-intervention assessment (T2), immediately following completion of the intervention
  Acceptability will be assessed at post-intervention (T2) using a structured 7-item survey evaluating perceived relevance, helpfulness, usability, satisfaction, and likelihood of recommending the intervention. Items are rated on a 5-point Likert scale (1 = strongly disagree/not helpful to 5 = strongly agree/very helpful).
  Metric: Number of participants rating items as 4 or 5 ÷ total number of respondents Unit of Measure: Percentage (%) of participants endorsing the acceptability threshold Benchmark: ≥ 80% of participants rate the intervention as helpful or very helpful (scores 4-5).
Qualitative Acceptability Feedback (Acceptability) | At the post-intervention assessment (T2), immediately following completion
  Qualitative acceptability will be assessed using open-ended questions examining perceived benefits, challenges, and recommendations for improvement of the HRVB intervention.
  Metric: Thematic saturation and frequency of key themes Unit of Measure: Narrative themes categorized as benefits, barriers, and recommendations Benchmark: Identification of actionable themes supporting feasibility and refinement of implementation.

SECONDARY OUTCOMES:
Perceived Sress | Baseline (T1) and 3 weeks after baseline (T2)
  Perceived stress will be measured using the 10-item Perceived Stress Scale (PSS-10), a validated self-report questionnaire that assesses the degree to which individuals perceive their lives as unpredictable, uncontrollable, and overwhelming during the past month. Higher scores indicate greater perceived stress.
Perceived Affect | Baseline (T1) and 3 weeks after baseline (T2)
  Affect will be measured using the Positive and Negative Affect Schedule (PANAS-SF, 20 items), a validated self-report measure that assesses the extent of positive affect (e.g., enthusiasm, alertness) and negative affect (e.g., distress, irritability) experienced over a specified time period. Higher scores indicate greater levels of the respective affective state. In addition, affect will be assessed through a brief daily diary using 12 PANAS-derived items to capture day-to-day fluctuations in positive and negative affect, providing a more nuanced understanding of affect over the 3-week study period.
Perceived difficulties in emotional regulation | Baseline (T1) and 3 weeks after baseline (T2)
  Perceived difficulties in emotional regulation will be measured using the Difficulties in Emotion Regulation Scale-Short Form (DERS-16), which is a validated self-report instrument that assesses global impairments in emotion regulation across multiple domains. It evaluates the frequency with which individuals experience problems such as heightened emotional reactivity, nonacceptance of emotional responses, difficulties maintaining goal-directed behavior when distressed, challenges controlling impulses during negative affect, and limited perceived access to effective emotion regulation strategies. Higher total scores reflect greater overall difficulty in regulating emotions.
Craving for illicit opioids | Baseline (T1) and 3 weeks after baseline (T2)
  Cravings for illicit opioids will be measured using the Obsessive Compulsive Drug Use Scale (OCDUS). This tool will be used to assess craving severity, capturing obsessive thoughts about substance use, compulsive urges, and perceived control over craving-related cognitions and behaviors. Higher scores indicate greater craving intensity and preoccupation with drug use. In addition, craving will be monitored through a brief daily diary item assessing subjective craving severity, allowing examination of day-to-day fluctuations and temporal patterns in craving experiences across the study period.
Perceived social support | Baseline (T1) and 3 weeks after baseline (T2)
  Perceived social support will be measured using The Multidimensional Scale of Perceived Social Support (MSPSS), which is a validated self-report instrument that assesses perceived adequacy of social support from three primary sources: family, friends, and significant others. It evaluates individuals' subjective sense of being valued, understood, and supported emotionally and practically by their social networks. Higher scores indicate greater perceived availability and quality of social support across these domains.
Self-efficacy to resist substance use | Baseline (T1) and 3 weeks after baseline (T2)
  The Drug-Taking Confidence Questionnaire-8 (DTCQ-8) is a brief, validated self-report measure of self-efficacy to resist substance use across high-risk situations. It assesses an individual's perceived confidence in their ability to refrain from using drugs when experiencing common triggers such as negative emotions, social pressure, craving, or interpersonal conflict. Higher scores indicate greater confidence in resisting drug use and a lower likelihood of relapse in these situations.
Autonomic regulation | Baseline (T1) and 3 weeks after baseline (T2)
  Heart rate variability (HRV) metrics, including SDNN, RMSSD, mean heart rate, mean interbeat interval (IBI), total power, LF, HF, and LF/HF ratio, will be used as objective indicators of autonomic nervous system functioning, reflecting overall variability, parasympathetic activity, and sympathetic-parasympathetic balance. In addition, normalized coherence scores from daily HeartMath Inner Balance practice will assess the degree of physiological synchronization and autonomic efficiency. Together, these measures provide complementary indices of autonomic regulation, stress resilience, and emotional regulation capacity, with higher variability and coherence generally indicating healthier autonomic functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States